CLINICAL TRIAL: NCT00184769
Title: Open Randomized Trial Examining the Growth and Safety Effects of Treatment With Recombinant Growth Hormone on Infants Aged 1 to 2 Years With Growth Retardation Secondary to Chronic Renal Insufficiency
Brief Title: Growth Hormone Treatment in Infants Aged 1 to 2 Years With Chronic Renal Insufficiency (CRI) and Growth Retardation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHCRF/E/2
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Chronic Kidney Disease; Chronic Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Europe. Objective(s): To evaluate the effect of human growth hormone on infants aged 1 to 2 years with chronic renal insufficiency (CRI) and growth retardation despite an adequate dietary intake.

Trial Design: This is an open, parallel group clinical trial with a duration of one year, in which period 50% of patients will receive GH treatment and the other 50% will act as a control group, without treatment.

Trial Population: The trial will involve a total of 16 infants aged from 12±3 to 24 months suffering chronic renal insufficiency (Glomerular Filtration Rate less than 60 ml/min/1.73 m2), and growth failure and undergoing conservative treatment or peritoneal dialysis. Include the key inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be infants of both sexes aged 12 ± 3 months with chronic renal insufficiency and growth retardation.
* To be included in the trial, patients must meet all of the following inclusion criteria a.)-c.):
* a.) Male or female infants with a chronological age of 12 ± 3 months
* b.) Chronic renal insufficiency with Glomerular Filtration Rate less than 60 ml/min./1.73m2, according to the method used routinely in each participating center
* c.) Growth retardation documented at the start of the trial, according to the following criteria: Length less than -2 SDS by chronological age and sex and linear growth velocity <P50 according to the Hernández standards and to Lubchenko in the case of infants born prematurely (<37 weeks)
* Conservative treatment or chronic peritoneal dialysis
* Euthyroid
* The parent or guardian must give informed consent to the child's participation in the study before any trial related activities. Trial related activities are any procedures that would not have been performed during the normal management of the subject
* Optimal nutritional management criteria met
* Appropriate metabolic control for severe hyperparathyroidism, hydroelectrolyte balance, acid-base balance and calcium-phosphorus balance

Exclusion Criteria:

* Any primary endocrinological disorder and severe renal osteodystrophy.Other causes, apart from CRI, giving rise to growth retardation.Hydrocephalus.
* Known or suspected allergy to the trial product or related products.
* Treatment with corticosteroids within the last six months.
* Renal disease due to the Fanconi syndrome or to oxalosis (except if not under dialysis).
* Known or suspected malignancy.

Ages: 9 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 1998-01-29 (Actual); Primary Completion 2005-12-21 (Actual); Study Completion 2005-12-21 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of growth hormone on infants aged 1 to 2 years with CRI and growth retardation growth retardation despite an adequate dietary intake | after 1 year of treatment

SECONDARY OUTCOMES:
Secondary objectives are to assess the safety of rhGH treatment in these infants. Safety assessment will include evaluation of renal function, Bone, IGF-I, IGFBP3 and psychological development

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (17):
- Portugal (3):
  - Novo Nordisk Investigational Site, Coimbra
  - Novo Nordisk Investigational Site, Lisbon
  - Novo Nordisk Investigational Site, Porto
- Spain (14):
  - Novo Nordisk Investigational Site, Badajoz
  - Novo Nordisk Investigational Site, Barakaldo
  - Novo Nordisk Investigational Site, Esplugues Llobregat
  - Novo Nordisk Investigational Site, Lugo
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Oviedo
  - Novo Nordisk Investigational Site, Pamplona
  - Novo Nordisk Investigational Site, San Sebastián
  - Novo Nordisk Investigational Site, Santa Cruz de Tenerife
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Zaragoza

REFERENCES:
- [Derived] Santos F, Moreno ML, Neto A, Ariceta G, Vara J, Alonso A, Bueno A, Afonso AC, Correia AJ, Muley R, Barrios V, Gomez C, Argente J. Improvement in growth after 1 year of growth hormone therapy in well-nourished infants with growth retardation secondary to chronic renal failure: results of a multicenter, controlled, randomized, open clinical trial. Clin J Am Soc Nephrol. 2010 Jul;5(7):1190-7. doi: 10.2215/CJN.07791109. Epub 2010 Jun 3. PMID 20522533
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com